CLINICAL TRIAL: NCT05941078
Title: An International Classification of Functioning, Disability and Health (ICF)-Based Post-stroke Program for Meeting Activity and Participation Needs in Patients
Brief Title: ICF Activity and Participation Needs in Post-stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The Hong Kong Society for Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PolyU RS ICF01
Record Dates: First submitted 2023-06-20; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-06

CONDITIONS: Stroke
Keywords: ICF; Stroke rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICF-based post-stroke rehabilitation program group (Experimental): The ICF-PSRP based on the ICF Core Set for Stroke targeted to facilitate patients' functional improvement, and community and social reintegration. Duration of the ICF-PSRP was eight or 12 weeks, comprising of 30 or 48 two-hour sessions depending on the patients' needs and progress.
  Interventions: Behavioral: ICF-based post-stroke rehabilitation program

INTERVENTIONS:
Behavioral: ICF-based post-stroke rehabilitation program — Patients completed an intake interview with a case therapist for an initial assessment and setting of personal treatment goals. The therapist assisted the patient with setting goals that were related to their life roles and functional gaps in terms of body function and activity and participation. Patients' personalized treatment plans were composed in case conferences. The treatment program contents were organized as ICF-based body function and activity and participation intervention modules. Each of the occupational therapy, physiotherapy, and speech therapy disciplines set the aims and developed the training contents, intensities, durations, and upgrading and completion criteria.

SUMMARY:
Stroke is regarded as one of the leading causes of adult mortality and disability. Conventional rehabilitation programs for post-stroke patients focus on the augmentation of body functions. Their service delivery models are mostly operationalized according to the individual discipline's knowledge domain and practices. The International Classification of Functioning, Disability and Health (ICF) model provides a comprehensive framework which places focus on patients' activity and participation. It also emphasizes cross-disciplinary integration of service provision, patient-centred approach and personalization of treatment aims. This study is aimed to investigate how the ICF model can be integrated into the planning and implementation of personalized post-stroke programs, and evaluate the program's effectiveness in fulfilling the activity and participation needs of patients.

DETAILED DESCRIPTION:
Stroke is a neurological disease and is regarded as one of the leading causes of adult mortality and disability. Post-stroke rehabilitation to promote functional recovery is important to restitute the brain tissue to relearn and compensate for the lost functions. Early rehabilitation to enhance neuroplasticity within three to six months of post-stroke is recommended to reduce neurological deficits caused by stroke. Promising stroke rehabilitation interventions to tackle mobility and cognitive impairments include fitness training, upper and lower extremity interventions, and reminiscence therapy.

The ICF model is proposed by the World Health Organization to describe health and health-related domains. It was developed based on the biopsychosocial model. Within the model, disability and functioning are identified as difficulties in 1) body functions and structure; 2) activity; and 3) participation. They are affected by the interaction between health conditions and contextual factors. The former is different diseases, disorders and injuries, while the latter consists of environmental factors and personal factors. The ICF model has been widely applied in assessment, treatment and evaluation in various disciplines. On top of the ICF model, there is a related neurorehabilitation process framed by ICF which makes up four steps. The first step is the assessment to understand the diagnosis and consequences of the current health condition of an individual. Followed by the goal-setting part to formulate short-term or long-term rehabilitation plans for patients' perspective. These two steps will inform the therapists of an ICF rehabilitation plan with corresponding ICF codes to describe patients' health conditions. The third step is to launch appropriate interventions based on the ICF rehabilitation plan, and the final step is the outcome measurements to review the appropriateness of interventions. Yet, a similar process has seldom been applied in post-stroke rehabilitation to guide the treatment program.

This project aims to investigate how the ICF model can be integrated into planning and implementation of an ICF-based post-stroke rehabilitation program (ICF-PSRP), and evaluate the program's effectiveness on fulfilling the activity and participation needs of patients.

ELIGIBILITY:
Inclusion Criteria:

1. had a diagnosis of stroke with an onset no more than 24 months,
2. were medically stable,
3. were able to transfer or walk with no more than one item of assistance, and
4. were able to tolerate at least 2 hours of active rehabilitation treatment.

Exclusion criteria:

1. Participants with neurological disabilities other than the stroke condition.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Modified Barthel Index | Baseline
  It measures the level of self-care management activities. Scores for the bladder, bowel, ambulation (indoor walking), stairs, dressing, feeding and on and off toilet items range from 0 to 10; transfer (bed mobility, sitting and floor), ambulation (outdoor walking), personal hygiene and bathing items range from 0 to 5. A higher score in each item indicates a better independence level, and vice versa for the dependence level on caregivers.
Modified Barthel Index | Up to 12 weeks
  It measures the level of self-care management activities. Scores for the bladder, bowel, ambulation (indoor walking), stairs, dressing, feeding and on and off toilet items range from 0 to 10; transfer (bed mobility, sitting and floor), ambulation (outdoor walking), personal hygiene and bathing items range from 0 to 5. A higher score in each item indicates a better independence level, and vice versa for the dependence level on caregivers.
Lawton Instrumental Activities of Daily Living Scale | Baseline
  It measures the level of independent living. All items in the scale range from 0 to 3. A higher score in each item indicates a better independence level, and vice versa for the dependence level on caregivers.
Lawton Instrumental Activities of Daily Living Scale | Up to 12 weeks
  It measures the level of independent living. All items in the scale range from 0 to 3. A higher score in each item indicates a better independence level, and vice versa for the dependence level on caregivers.
Elderly Mobility Scale | Baseline
  It measures the mobility level. The lying to sitting and sitting to lying items range from 0 to 2. The functional reach item ranges from 0 to 4. Other items, including sit to stand, stand, gait and time walk, range from 0 to 3. A higher score in each item indicates a better independence level, and vice versa for the dependence level on caregivers.
Elderly Mobility Scale | Up to 12 weeks
  It measures the mobility level. The lying to sitting and sitting to lying items range from 0 to 2. The functional reach item ranges from 0 to 4. Other items, including sit to stand, stand, gait and time walk, range from 0 to 3. A higher score in each item indicates a better independence level, and vice versa for the dependence level on caregivers.
Therapy Outcome Measure | Baseline
  It assesses patients' abilities and difficulties in terms of their impairment, activity, participation, and well-being in expressive and receptive language abilities. All items range from 0 to 5. A lower score reflects severely impaired language abilities, while scores close to 5 indicate less impaired or no impairment in language abilities.
Therapy Outcome Measure | Up to 12 weeks
  It assesses patients' abilities and difficulties in terms of their impairment, activity, participation, and well-being in expressive and receptive language abilities. All items range from 0 to 5. A lower score reflects severely impaired language abilities, while scores close to 5 indicate less impaired or no impairment in language abilities.
Manual Muscle Testing - Lower Extremity | Baseline
  It measures lower extremity muscle strength impairments. The score ranges from 0 to 5. A lower score indicates a trend of weak or no movements detected on the lower extremity. A higher score indicates a trend of slight decline or no impairments in muscle contraction under full resistance.
Manual Muscle Testing - Lower Extremity | Up to 12 weeks
  It measures lower extremity muscle strength impairments. The score ranges from 0 to 5. A lower score indicates a trend of weak or no movements detected on the lower extremity. A higher score indicates a trend of slight decline or no impairments in muscle contraction under full resistance.
Functional Test for the Hemiplegic Upper Extremity | Baseline
  It measures the recovery of the hemiplegic upper extremity. The score ranges from level 1 to level 7 based on Brunnstrom's developmental stages of stroke recovery. A lower level reveals the severe impairment of the upper extremity to perform simple hand movements. A higher level indicates less or no impairments on the upper extremity to perform fine hand functional tasks.
Functional Test for the Hemiplegic Upper Extremity | Up to 12 weeks
  It measures the recovery of the hemiplegic upper extremity. The score ranges from level 1 to level 7 based on Brunnstrom's developmental stages of stroke recovery. A lower level reveals the severe impairment of the upper extremity to perform simple hand movements. A higher level indicates less or no impairments on the upper extremity to perform fine hand functional tasks.
Oxford Cognitive Screen | Baseline
  It measures stroke-induced cognitive disabilities. Areas include attention (score ranges from 0 to 63), memory (score ranges from 0 to 12), language (score ranges from 0 to 22), praxis (score ranges from 0 to 12) and number (score ranges from 0 to 4). A higher score indicates fewer impairments in the specific area, and vice versa for a lower score in the specific area.
Oxford Cognitive Screen | Up to 12 weeks
  It measures stroke-induced cognitive disabilities. Areas include attention (score ranges from 0 to 63), memory (score ranges from 0 to 12), language (score ranges from 0 to 22), praxis (score ranges from 0 to 12) and number (score ranges from 0 to 4). A higher score indicates fewer impairments in the specific area, and vice versa for a lower score in the specific area.

SECONDARY OUTCOMES:
Goal Attainment Scale | Baseline
  It enables patients to set individualised achievable goals at the beginning of the program. The score ranges from -2 to +2. All patients begin at the level of -2. A zero score indicates patients' improvements to reach their goal(s). A +2 score indicates an out-of-expectation improvement in the program.
Stroke Specific Quality of Life Scale | Baseline
  It measures post-stroke patients' health-related quality of life with good internal consistency. All items range from 1 to 5. A lower item score implies a disagreement or requirement of total help from patients' perspectives, and vice versa for a higher item score. The same interpretation applies to the sum of scores.
Stroke Specific Quality of Life Scale | Up to 12 weeks
  It measures post-stroke patients' health-related quality of life with good internal consistency. All items range from 1 to 5. A lower item score implies a disagreement or requirement of total help from patients' perspectives, and vice versa for a higher item score. The same interpretation applies to the sum of scores.

CONTACTS AND LOCATIONS:
Overall Officials: Che Hin Chetwyn Chan, PhD, Study Chair — The Education University of Hong Kong
Locations (1):
- The Hong Kong Society for Rehabilitation Cheng Tak Yim Day Rehabilitation and Care Centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The collected data, such as treatment goal contents, assessment results and demographic variables, may reveal participants' identities. Further, participants were not informed about sharing their information with parties other than the research team and rehabilitation centre.

REFERENCES:
- [Derived] Wong MN, Cheung MK, Ng YM, Yuan HL, Lam BY, Fu SN, Chan CCH. International Classification of Functioning, Disability, and Health-based rehabilitation program promotes activity and participation of post-stroke patients. Front Neurol. 2023 Nov 3;14:1235500. doi: 10.3389/fneur.2023.1235500. eCollection 2023. PMID 38020626